CLINICAL TRIAL: NCT07287956
Title: The Use of Adjunct Oxygen High-Level Laser Therapy on the Clinical and Microbiological Outcomes of Peri-implant Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20240239
Record Dates: First submitted 2025-08-26; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-08

CONDITIONS: Peri-Implantitis and Peri-implant Mucositis
Keywords: photodynamic therapy; hydrogen peroxide; oxygen high-level laser therapy; microbiology; modified photodynamic therapy; diode laser
MeSH Terms: conditions — Peri-Implantitis | interventions — Lasers, Semiconductor; Hydrogen Peroxide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Diode laser and hydrogen peroxide (Active Comparator): The dental implant will receive treatment using diode laser and hydrogen peroxide following mechanical debridement.
  Interventions: Combination Product: Oxygen high-level laser therapy (Diode laser and hydrogen peroxide)
- Diode laser (Active Comparator): The dental implant will receive treatment using diode laser following mechanical debridement.
  Interventions: Device: Diode laser therapy

INTERVENTIONS:
Combination Product: Oxygen high-level laser therapy (Diode laser and hydrogen peroxide) — After mechanical debridement of the affected dental implant, a 3% hydrogen peroxide solution will be applied to the peri-implant pocket. This will be followed by irradiation using a diode laser at 940nm wavelength, applied for 60 seconds per site. The intervention will be performed in a single treatment session.
  Arms: Diode laser and hydrogen peroxide
Device: Diode laser therapy — After mechanical debridement of the affected dental implant, irradiation using a diode laser at 940nm wavelength, applied for 60 seconds per site will be performed. This intervention will be administered in a single treatment session.
  Arms: Diode laser

SUMMARY:
The goal of this clinical trial is to learn whether using a special light-activated treatment called photodynamic therapy, or more specifically, its modified version called oxygen high-level laser therapy, using a high-powered diode laser along with 3% hydrogen peroxide, can improve gum health around dental implants. It tests whether adding this to regular cleaning treatments could reduce harmful bacteria and support better healing. The aim is to determine whether a specific protocol is an effective way to treat infections around dental implants.

Participants in the study will receive two types of treatment on different dental implants:

* One implant will be treated with the oxygen high-level laser therapy using diode laser and hydrogen peroxide after mechanical cleaning.
* The other implant will receive diode laser therapy without hydrogen peroxide after mechanical cleaning.

Researchers will compare how the gums respond to each treatment, looking at signs such as inflammation, and determine whether the number of harmful bacteria has been reduced at three time points.

DETAILED DESCRIPTION:
Participants attending with at least two non-adjacent dental implants diagnosed with peri-implant disease (peri-implant mucositis and peri-implantitis) will be enrolled in the study. All patients included will be examined, and periodontal chartings will be obtained using a PCPUNC 15 probe. After routine phase one therapy (mechanical debridement using carbon-coated curettes on dental implants and ultrasonic scaling on the rest of the dentition), implant pocket irrigation using normal saline will be performed in both groups. Following irrigation using normal saline, implant pockets will be irrigated with 3% hydrogen peroxide, left in place for 2 minutes, and then irradiated with a 940nm diode laser (2.5W power, high frequency, 10 KHz, power average 0.5 W, fluency 25,000 J/cm2, 416.66 J/cm2 per second [Rey Protocol]) for 60 s per site in the test group. Control groups will receive mechanical debridement and diode laser treatment alone without the use of hydrogen peroxide.

Baseline clinical parameters will be measured at the initial visit and compared to post-treatment results at 6 weeks and 3 months. The clinical parameters to be evaluated include probing pocket depth, gingival index, plaque index, bleeding on probing, and suppuration.

In addition, microbiological parameters (bacterial count) using quantitative real-time polymerase chain reaction (qPCR) analysis will be determined from subgingival plaque samples using sterile paper points before and after treatment of both groups left in place for 30 seconds. Supragingival plaque is to be removed, and microbiological samples are to be taken before any measurements and/or non-surgical periodontal therapy (NSPT) from the deepest peri-implant pockets (sites are to be isolated with cotton rolls and gently air dried to avoid contamination with saliva). Immediately following treatment, a second swab will be taken from the implant surface using the same procedure discussed previously. Further samples will be collected at 6 week and 3-month follow-ups and processed.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older.
* Patients diagnosed with peri-implant disease (peri-implant mucositis or peri-implantitis) according to the 2017 World Workshop criteria in at least two non-adjacent, single-crown, bone-level dental implants.
* Patients that have not undergone periodontal treatment and/or were prescribed antibiotics in the last three months prior to initial visit.
* Patients with a healthy periodontal status
* At least 1 year of functional implants.
* Non-Smokers.

Exclusion Criteria:

* Immunocompromised patients.
* Pregnancy or breastfeeding.
* Known allergies to any materials used in the study.
* Patients classified as ASA Physical Status ≥ III.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Probing Pocket Depth | From enrollment to the end of follow-ups at 3 months.
  Probing pocket depth (PPD): The distance from the gum margin to the bottom of the pocket around a tooth or implant using a periodontal probe.
  Measurements were taken using PCPUNC 15 periodontal probe inserted parallel to the long axis of the implant until soft resistance was felt. Six sites per implant were recorded (mesiobuccal, mid-buccal, distobuccal, mesio-oral, mid-oral, disto-oral), and mean values were calculated. Higher values indicate deeper pockets and greater inflammation.
  Unit of Measure: millimeters (mm)
Bleeding on Probing | From enrollment to the end of follow-ups at 3 months
  Bleeding on Probing (BOP): Percentage of sites exhibiting bleeding upon gentle probing around a tooth or implant using a periodontal probe. Each site was scored as bleeding (yes) or not bleeding (no) within 30 seconds after probing.
  The percentage of bleeding sites was calculated as:
  (number of bleeding sites ÷ total sites) × 100.
  Higher percentages indicate greater inflammatory response. Unit of Measure: Percentage (%)
Gingival Index | From enrollment to the end of follow-ups at 3 months
  Gingival index: A clinical measure used to assess the severity of gingival inflammation. It is based on the color, consistency, and bleeding of the gums when gently probed.
  The scale ranges from 0 to 3, where:
  0 = normal gingiva (no inflammation)
  1. = mild inflammation (slight color change, no bleeding on probing)
  2. = moderate inflammation (redness, edema, bleeding on probing)
  3. = severe inflammation (marked redness, ulceration, spontaneous bleeding)
  Higher scores indicate more severe inflammation. Unit of Measure: Units on a scale (0-3)
Plaque Index | From enrollment to the end of follow-ups at 3 months
  Plaque index: A scoring system used to measure the amount of dental plaque on the teeth or implants.
  The scale ranges from 0 to 3, where:
  0 = no plaque detected
  1. = plaque only detectable by probe
  2. = visible plaque
  3. = abundant plaque accumulation
  Higher scores indicate greater plaque accumulation. Unit of Measure: Units on a scale (0-3)

SECONDARY OUTCOMES:
Bacterial Load of Peri-Implant Pathogens (qPCR) | From enrollment to the end of follow-ups at 3 months.
  Quantitative measurement of target peri-implant bacteria (Porphyromonas gingivalis, Tannerella forsythia, Aggregatibacter actinomycetemcomitans, Fusobacterium nucleatum, Streptococcus mutans) using qPCR.
  Unit of Measure: Copies per microliter (copies/µL)
Suppuration | From enrollment to the end of follow-ups at 3 months
  Suppuration was assessed by applying gentle pressure with a periodontal probe at six peri-implant sites.
  Any detectable exudate or pus was recorded as "present"; absence of exudate was recorded as "absent." Presence of suppuration indicates active infection.
  Unit of Measure: Presence/Absence (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Rola Alhabashneh, Study Chair — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and Technology, Irbid, Alabama, Jordan

IPD SHARING:
Plan to Share IPD: Undecided
Privacy and confidentiality of patients.